CLINICAL TRIAL: NCT01838395
Title: A Phase IIa, Multicenter, Open-Label Study Designed to Evaluate the Safety and Efficacy of Escalating Doses of BL-8040 in Adult Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Brief Title: Phase IIa Study Evaluating Safety and Efficacy of BL-8040 in Relapsed/Refractory AML Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-8040.01
Record Dates: First submitted 2013-04-14; First posted 2013-04-24 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; 4-fluorobenzoyl-TN-14003

STUDY DESIGN:
Intervention Model Description: The study (Part 1) will include escalating dose groups and be considered the 'escalation phase'. Five potential dose levels will be investigated starting at dose level 1. Patients will be accrued in a conventional 3+3 design. Applying this study design, the first cohort of 3 patients will be treated at dose level 1 and evaluated for dose escalation.
  Dose escalation will be permitted until the Maximum Tolerated Dose (MTD) is established and protocol specific stopping rules for toxicity are met. If no MTD is reached, dose escalation will continue up to dose level 5 (1.5 mg/kg).
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- BL-8040 0.5mg/kg + Ara-C 1.5 or 3 g/m2/d per dose (based on age) (Experimental): Arm 1: Participants will be dosed with SC injections of BL-8040 over two days followed by concurrent administration of 0.5 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) during 5 days.
  Interventions: Drug: Ara-C; Drug: BL-8040
- BL-8040 0.75mg/kg + Ara-C 1.5 or 3 g/m2/d (based on age) (Experimental): Arm 2: Participants will be dosed with SC injections of BL-8040 over two days followed by concurrent administration of 0.75 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) during 5 days.
  Interventions: Drug: Ara-C; Drug: BL-8040
- BL-8040 1.0mg/kg + Ara-C 1.5 or 3 g/m2/d (based on age) (Experimental): Arm 3: Participants will be dosed with SC injections of BL-8040 over two days followed by concurrent administration of 1 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) during 5 days.
  Interventions: Drug: Ara-C; Drug: BL-8040
- BL-8040 1.25mg/kg + Ara-C 1.5 or 3 g/m2/d (based on age) (Experimental): Arm 4: Participants will be dosed with SC injections of BL-8040 over two days followed by concurrent administration of 1.25 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) during 5 days.
  Interventions: Drug: Ara-C; Drug: BL-8040
- BL-8040 1.5mg/kg + Ara-C 1.5 or 3 g/m2/d (based on age) (Experimental): Arm 5: Participants will be dosed with SC injections of BL-8040 over two days followed by concurrent administration of 1.5 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) during 5 days.
  Interventions: Drug: Ara-C; Drug: BL-8040
- BL-8040 2mg/kg + Ara-C 1.5 or 3 g/m2/d (based on age) (Experimental): Arm 6: Participants will be dosed with SC injections of BL-8040 over two days followed by concurrent administration of 2 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) during 5 days.
  Interventions: Drug: Ara-C; Drug: BL-8040

INTERVENTIONS:
Drug: Ara-C — IV (intravenous administration)
  Other Names: Cytarabine
Drug: BL-8040 — SC (subcutaneous injection)

SUMMARY:
A study is designed to assess if BL-8040 in combination with cytarabine (Ara-C) can help controlling the disease in patients with Acute Myeloid Leukemia (AML) that have relapsed or did not respond adequately to previous treatment. The safety of the study drug combination will also be studied.

DETAILED DESCRIPTION:
Open-label, multicenter, Phase IIa, dose escalating study in subjects with relapsed/refractory AML, defined according to WHO criteria, including subjects who failed chemotherapy only and those who failed previous Autologous Stem Cell Transplantation (ASCT)/ Allogeneic Stem Cell Transplantation (AlloSCT), provided at least 6 months have passed from transplant.

Eligible subjects will receive subcutaneous (SC) injections of BL-8040 ("monotherapy period") over two days (one injection per day) followed by concurrent administration of BL-8040 with standard salvage chemotherapy ("combined period") over 5 days. During the "combined period," BL-8040 will be administered 4 hours prior to chemotherapy. The chemotherapy will consist of cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age), administered intravenously (IV) over 3 hours, for 5 days and will not be escalated.

The first part of the study (Part 1) will include escalating dose groups and be considered the 'escalation phase'. Six potential dose levels will be investigated starting at dose level 1. Patients will be accrued in a conventional 3+3 design. Applying this study design, the first cohort of 3 patients will be treated at dose level 1 and evaluated for dose escalation.

At the discretion of the Sponsor, additional subjects may be enrolled into a selected dose group to confirm safety and efficacy for selected dose. the portion of this study is considered expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women subjects aged 18 to 75, inclusive.
2. Confirmed diagnosis of relapsed/refractory AML (WHO criteria) Refractory subjects, up to second consecutive salvage . Relapsed subjects including first and second relapse.
3. AML relapse > 6 months since autologous or allogeneic stem cell transplantation, provided they are in first or second relapse and:

   No active graft-versus-host disease (GVHD > grade 1). No treatment with high dose steroids for GVHD (up to 20 mg Prednisolone or equivalent, Appendix G). No treatment with immunosuppressive drugs with the exception of low dose cyclosporine and tacrolimus (blood levels of 0.5-0.6 µg/mL).
4. Clinical laboratory values should be as follows:

   White Blood Cells (WBC) < 30,000/mL Blasts in Peripheral Blood (PB) ≤ 20,000. Treatment with Hydroxyurea is permitted up to 24 hrs prior to BL-8040 administration to achieve blast counts < 20,000 prior to enrollment. Creatinine < 1.3 mg/dL; if Creatinine is > 1 mg/dL the Creatinine clearance should be > 40 mL/min as calculated using the Cockcroft-Gault formula.
5. Women of childbearing potential and all men must agree to use an approved form of contraception (e.g. oral, transdermal patch, implanted contraceptives, intrauterine device, diaphragm, condom, abstinence or surgical sterility) prior to study entry and for the duration of study participation through 30 days after the last dose of BL-8040. Confirmation that female subjects are not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
6. Subject is able and willing to comply with the requirements of the protocol.
7. Subject is able to voluntarily provide written informed consent.

Exclusion Criteria:

1. Administration of conventional chemotherapy within 2 weeks of enrollment date. In the event that subjects have received chemotherapy > 2 weeks from the date of enrollment, they may be included provided they have recovered from the associated non-hematological toxicities to ≤ grade 1.
2. Life expectancy of ≤ 2 months.
3. Known allergy or hypersensitivity to any of the test compounds, materials or contraindication to test product.
4. Use of investigational device or agents within 2 weeks of enrollment date.
5. Low Performance Status (ECOG > 2; Appendix E).
6. O2 saturation < 92% (on room air), evidence of Tumor Lysis Syndrome (TLS) > grade 2 (according to the Cairo-Bishop criteria (3)) or leukostasis (2).
7. Abnormal liver function tests:

   Serum aspartate transaminase (AST/SGOT) or alanine transaminase ( Alanine Transaminase (ALT)/Serum Glutamic Pyruvic Transaminase (SGPT)) 2 x upper limit of normal (ULN).

   Serum bilirubin. Total bilirubin > 2.0 mg/dL (34 µmol/L), conjugated bilirubin > 0.8 mg/dL.
8. Left ventricular ejection fraction < 40 %.
9. History of myocardial infarction or cerebrovascular accident within 6 months of enrollment date.
10. Presence of active, uncontrolled infection.
11. Known central nervous system disease (e.g., Alzheimer's disease).
12. Acute promyelocytic leukemia.
13. Exposure to high dose Ara-C within 6 months of enrollment.
14. Subject has concurrent, uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place him/her at unacceptable risk, including, but not limited to:

    Subject has been diagnosed or treated for another malignancy within 3 years of enrolment, except in situ malignancy, or low-risk prostate, skin or cervix cancer after curative therapy A co-morbid condition which, in the view of the Investigators, renders the subject at high risk from treatment complications.
15. Female subjects who are pregnant or breastfeeding.
16. Prior clinically significant grade 3-4 non-hematological toxicity to high dose Ara-C or grade ≥ 2 of neurological toxicity.
17. Seropositive for HIV antibodies (HIV1 and HIV2), Hepatitis C antibody (Hep C Ab) or a Hepatitis B carrier (positive for Hepatitis B surface antigen [HBsAg]).
18. Unable to comply with study requirements in the opinion of the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Aharon, MD, Study Chair — BioLineRx, Ltd.
Locations (10):
- United States (5):
  - Mayo Clinic, Jacksonville, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included 6 escalating dose groups
  The decision to proceed to the next dose level was made by an independent Data Monitoring Committee (DMC) after review of the relevant safety data. At the discretion of the Sponsor, additional subjects could be enrolled into a selected dose group to confirm the safety, efficacy and pharmacokinetic (PK) profile for the selected dose.
Groups:
- Period 1: BL-8040 0.5 mg/kg + Ara-C: Participants were dosed with SC injections of 0.5 mg/kg BL-8040 over two days followed by concurrent administration of 0.5 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 2: BL-8040 0.75 mg/kg + Ara-C: Participants were dosed with SC injections of 0.75 mg/kg BL-8040 over two days followed by concurrent administration of 0.75 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 3: BL-8040 1.0 mg/kg + Ara-C: Participants were dosed with SC injections of 1.0 mg/kg BL-8040 over two days followed by concurrent administration of 1.0 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 4: BL-8040 1.25 mg/kg + Ara-C: Participants were dosed with SC injections of 1.25 mg/kg BL-8040 over two days followed by concurrent administration of 1.25 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 5 & Expansion Phase: BL-8040 1.5 mg/kg + Ara-C: Participants were dosed with SC injections of 1.5 mg/kg BL-8040 over two days followed by concurrent administration of 1.5 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 6: BL-8040 2.0 mg/kg + Ara-C: Participants were dosed with SC injections of 2.0 mg/kg BL-8040 over two days followed by concurrent administration of 2.0 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
Period: Overall Study
Arm/Group | Period 1: BL-8040 0.5 mg/kg + Ara-C | Period 2: BL-8040 0.75 mg/kg + Ara-C | Period 3: BL-8040 1.0 mg/kg + Ara-C | Period 4: BL-8040 1.25 mg/kg + Ara-C | Period 5 & Expansion Phase: BL-8040 1.5 mg/kg + Ara-C | Period 6: BL-8040 2.0 mg/kg + Ara-C
Started | 3 | 3 | 6 | 4 | 23 | 3
Completed | 3 | 2 | 5 | 4 | 22 | 3
Not Completed | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — started conditioning regimen prior to hematopoietic stem cell transplant | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Period 1: 0.5 mg/kg BL-8040 + Ara-C: 0.5 mg/kg BL-8040 administration over two days followed by concurrent administration of 0.5 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 2: 0.75 mg/kg BL-8040 + Ara-C: 0.75 mg/kg BL-8040 administration over two days followed by concurrent administration of 0.75 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 3: 1.0 mg/kg BL-8040 + Ara-C: 1.0 mg/kg BL-8040 administration over two days followed by concurrent administration of 1.0 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 4: 1.25 mg/kg BL-8040 + Ara-C: 1.25 mg/kg BL-8040 administration over two days followed by concurrent administration of 1.25 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 5 & Expansion Phase: 1.5 mg/kg BL-8040 + Ara-C: 1.5 mg/kg BL-8040 administration over two days followed by concurrent administration of 1.5 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 6: 2.0 mg/kg BL-8040 + Ara-C: 2.0 mg/kg BL-8040 administration over two days followed by concurrent administration of 2.0 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Total: Total of all reporting groups
Arm/Group | Period 1: 0.5 mg/kg BL-8040 + Ara-C | Period 2: 0.75 mg/kg BL-8040 + Ara-C | Period 3: 1.0 mg/kg BL-8040 + Ara-C | Period 4: 1.25 mg/kg BL-8040 + Ara-C | Period 5 & Expansion Phase: 1.5 mg/kg BL-8040 + Ara-C | Period 6: 2.0 mg/kg BL-8040 + Ara-C | Total
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 23 | 3 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.5) | 62.0 (6.1) | 56.8 (10.9) | 62.3 (10.2) | 61.3 (8.8) | 52.3 (20.0) | 60.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 10 | 2 | 19
  Male | 1 | 2 | 4 | 2 | 13 | 1 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 6 | 4 | 20 | 2 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Number of participants with Adverse event affecting the safety and tolerability of BL-8040 + Ara-C by dose level (overall, dose limiting events, related Adverse Events (AEs), Serious Adverse Events (SAEs), related SAEs, AE by severity and death) Toxicity grade was assessed according to version V4.03 of NCI-CTCAE
Time Frame: Participants were followed for the duration of the hospital stay and the follow-up period, an expected average of 6 weeks.
Population: All patients who received at least one dose of BL-8040 were included in the analysis (ITT)
Measure: Count of Participants; unit: Participants
Groups:
- BL-8040 + Ara-C: Eligible subjects received subcutaneous (SC) injections of BL-8040 ("monotherapy period") over two days (one injection per day) followed by concurrent administration of BL-8040 with standard salvage chemotherapy ("combined period") over 5 days. During the "combined period," BL-8040 was be administered 4 hours prior to chemotherapy. The chemotherapy consisted of cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age), administered intravenously (IV) over 3 hours, for 5 days without escalation.
  Ara-C: IV
  BL-8040: SC
- Period 1: BL-8040 0.5 mg/kg + Ara-C: 0.5 mg/kg BL-8040 administration over two days followed by concurrent administration of 0.5 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 2: BL-8040 0.75 mg/kg + Ara-C: 0.75 mg/kg BL-8040 administration over two days followed by concurrent administration of 0.75 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days
- Period 3: BL-8040 1.0 mg/kg + Ara-C: 1.0 mg/kg BL-8040 administration over two days followed by concurrent administration of 1.0 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 4: BL-8040 1.25 mg/kg + Ara-C: 1.25 mg/kg BL-8040 administration over two days followed by concurrent administration of 1.25 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 5 & Expansion: BL-8040 1.5 mg/kg + Ara-C: 1.5 mg/kg BL-8040 administration over two days followed by concurrent administration of 1.5 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
- Period 6: BL-8040 2.0 mg/kg + Ara-C: 2.0 mg/kg BL-8040 administration over two days followed by concurrent administration of 2.0 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
Arm/Group | BL-8040 + Ara-C | Period 1: BL-8040 0.5 mg/kg + Ara-C | Period 2: BL-8040 0.75 mg/kg + Ara-C | Period 3: BL-8040 1.0 mg/kg + Ara-C | Period 4: BL-8040 1.25 mg/kg + Ara-C | Period 5 & Expansion: BL-8040 1.5 mg/kg + Ara-C | Period 6: BL-8040 2.0 mg/kg + Ara-C
Number analyzed (Participants) | 42 | 3 | 3 | 6 | 4 | 23 | 3
Participants
  Adverse event: Subjects with any adverse event (per patient) | 42 | 3 | 3 | 6 | 4 | 23 | 3
  Adverse event: Subjects with any dose-limiting event (per patient) | 3 | 0 | 0 | 0 | 0 | 3 | 0
  Adverse event: Subjects with any drug-related AE (Definite/Probable) | 35 | 1 | 3 | 4 | 4 | 20 | 3
  Adverse event: Subjects with any drug-related AE (Definite/Probable/Possible) | 40 | 2 | 3 | 5 | 4 | 23 | 3
  Adverse event: Subjects with any serious AE | 21 | 1 | 3 | 3 | 1 | 10 | 3
  Adverse event: Subjects with any serious AE also drug-related (Definite/Probable) | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Adverse event: Subjects with serious AE also drug-related (Definite/Probable/Possible) | 3 | 0 | 0 | 0 | 0 | 3 | 0
  Adverse event : Subjects with severe or life-threatening AE | 33 | 2 | 3 | 4 | 2 | 19 | 3
  Adverse event : Subjects with mild and/or moderate AE | 41 | 3 | 3 | 6 | 4 | 22 | 3
  Adverse event : Death | 2 | 0 | 0 | 1 | 1 | 0 | 0

2. Secondary Outcome: Response to Treatment by Dose
Description: Response rate as assessed at final bone marrow evaluation based on Cheson et al 2003 criteria.
  * CR defined as bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 10^9/L (1000/μL); platelet count >100 x 10^9/L (100,000/μL); independent of red cell transfusions
  * CRi defined as all CR criteria except for residual neutropenia (<1.0 x 10^9/L [1000/μL]) or thrombocytopenia (<100 x 10^9/L [100,000/μL])
  * Partial Response (PR) defined as all hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%
Time Frame: Final bone marrow evaluation - Between Day 20 and Day 44
Measure: Number; unit: participants
Groups:
- Period 5 & Expansion: BL-8040 1.5 mg/kg + Ara-C: Participants were dosed with SC injections of 1.5 mg/kg BL-8040 over two days followed by concurrent administration of 1.5 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days.
Arm/Group | Period 1: BL-8040 0.5 mg/kg + Ara-C | Period 2: BL-8040 0.75 mg/kg + Ara-C | Period 3: BL-8040 1.0 mg/kg + Ara-C | Period 4: BL-8040 1.25 mg/kg + Ara-C | Period 5 & Expansion: BL-8040 1.5 mg/kg + Ara-C | Period 6: BL-8040 2.0 mg/kg + Ara-C
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 23 | 3
participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 4 | 0
  Complete response with incomplete recovery (CRi) | 0 | 0 | 2 | 1 | 5 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 1 | 1
  Overall Response (CR+CRi+PR) | 0 | 0 | 2 | 1 | 10 | 1
  Complete Response (CR and CRi) | 0 | 0 | 2 | 1 | 9 | 0

3. Secondary Outcome: Apoptotic Effect
Description: Change in leukemic cell apoptosis in peripheral blood and bone marrow
Time Frame: Final evaluation - between Day 20 and Day 44
Population: Data were not collected
Arm/Group | Period 1: BL-8040 0.5 mg/kg + Ara-C | Period 2: BL-8040 0.75 mg/kg + Ara-C | Period 3: BL-8040 1.0 mg/kg + Ara-C | Period 4: BL-8040 1.25 mg/kg + Ara-C | Period 5 & Expansion Phase: BL-8040 1.5 mg/kg + Ara-C | Period 6: BL-8040 2.0 mg/kg + Ara-C
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Assessment of the Pharmacokinetic Profile of BL-8040 - t1/2 (h)
Description: Pharmacokinetics (PK) of BL-8040 after daily subcutaneous (SC) dosing for 2 days alone, followed by 5 days of combined administration of BL-8040 + Ara-C by dose level.
  Standard Deviation is reported for N ≥ 3 t1/2 (h): The time required for plasma concentration of a drug to decrease by 50%
Time Frame: Blood samples for the determination of BL-8040 were collected before dosing and at 0.25, 0.5, 1, 2, 4, 8, and 24 hours after BL-8040 administration on Day 1.
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Period 1: 0.5 mg/kg BL-8040 + Ara-C | Period 2: 0.75 mg/kg BL-8040 + Ara-C | Period 3: 1.0 mg/kg BL-8040 + Ara-C | Period 4: 1.25 mg/kg BL-8040 + Ara-C | Period 5 & Expansion Phase: 1.5 mg/kg BL-8040 + Ara-C | Period 6: 2.0 mg/kg BL-8040 + Ara-C
Number analyzed (Participants) | 1 | 3 | 5 | 4 | 18 | 3
hours | 1.23 | 1.50 (0.484) | 1.40 (0.336) | 2.06 (1.92) | 2.11 (1.57) | 2.67 (1.27)

5. Secondary Outcome: Assessment of the Pharmacokinetic Profile of BL-8040 - Tmax (h)
Description: Pharmacokinetics (PK) of BL-8040 after daily subcutaneous (SC) dosing for 2 days alone, followed by 5 days of combined administration of BL-8040 + Ara-C by dose level.
  Standard Deviation is reported for N ≥ 3 tmax (h): The time to peak concentration
Time Frame: as for outcome 4
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Period 1: 0.5 mg/kg BL-8040 + Ara-C | Period 2: 0.75 mg/kg BL-8040 + Ara-C | Period 3: 1.0 mg/kg BL-8040 + Ara-C | Period 4: 1.25 mg/kg BL-8040 + Ara-C | Period 5 & Expansion Phase: 1.5 mg/kg BL-8040 + Ara-C | Period 6: 2.0 mg/kg BL-8040 + Ara-C
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 19 | 3
hours | 0.833 (0.289) | 0.417 (0.144) | 0.792 (0.332) | 0.875 (0.250) | 0.618 (0.281) | 1 (0)

6. Secondary Outcome: Assessment of the Pharmacokinetic Profile of BL-8040 - Cmax (ng/mL)
Description: Pharmacokinetics (PK) of BL-8040 after daily subcutaneous (SC) dosing for 2 days alone, followed by 5 days of combined administration of BL-8040 + Ara-C by dose level.
  Standard Deviation is reported for N ≥ 3 Cmax is the highest concentration of a drug in the blood
Time Frame: as for outcome 4
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Period 1: 0.5 mg/kg BL-8040 + Ara-C | Period 2: 0.75 mg/kg BL-8040 + Ara-C | Period 3: 1.0 mg/kg BL-8040 + Ara-C | Period 4: 1.25 mg/kg BL-8040 + Ara-C | Period 5 & Expansion Phase: 1.5 mg/kg BL-8040 + Ara-C | Period 6: 2.0 mg/kg BL-8040 + Ara-C
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 19 | 3
ng/mL | 380 (33.6) | 376 (155) | 712 (277) | 1670 (522) | 1940 (803) | 4020 (1510)

7. Secondary Outcome: Assessment of the Pharmacokinetic Profile of BL-8040 - AUC0-t (h*ng/mL)
Description: Pharmacokinetics (PK) of BL-8040 after daily subcutaneous (SC) dosing for 2 days alone, followed by 5 days of combined administration of BL-8040 + Ara-C by dose level.
  Standard Deviation is reported for N ≥ 3 AUC0-t is the Area Under the Curve (AUC), definite integral of the concentration of a drug in blood as a function of time.
Time Frame: as for outcome 4
Population: PK Population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Period 1: 0.5 mg/kg BL-8040 + Ara-C | Period 2: 0.75 mg/kg BL-8040 + Ara-C | Period 3: 1.0 mg/kg BL-8040 + Ara-C | Period 4: 1.25 mg/kg BL-8040 + Ara-C | Period 5 & Expansion Phase: 1.5 mg/kg BL-8040 + Ara-C | Period 6: 2.0 mg/kg BL-8040 + Ara-C
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 19 | 3
h*ng/mL | 661 (55.3) | 792 (447) | 1390 (541) | 3020 (1340) | 3650 (1640) | 8340 (2290)

8. Secondary Outcome: Assessment of the Pharmacokinetic Profile of BL-8040 - AUC0-24 (h*ng/mL)
Description: Pharmacokinetics (PK) of BL-8040 after daily subcutaneous (SC) dosing for 2 days alone, followed by 5 days of combined administration of BL-8040 + Ara-C by dose level.
  Standard Deviation is reported for N ≥ 3 AUC0-24 is the Area Under the Curve (AUC), definite integral of the concentration of a drug in blood from time zero to 24 hours post dose.
Time Frame: as for outcome 4
Population: PK Population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Period 1: 0.5 mg/kg BL-8040 + Ara-C | Period 2: 0.75 mg/kg BL-8040 + Ara-C | Period 3: 1.0 mg/kg BL-8040 + Ara-C | Period 4: 1.25 mg/kg BL-8040 + Ara-C | Period 5 & Expansion Phase: 1.5 mg/kg BL-8040 + Ara-C | Period 6: 2.0 mg/kg BL-8040 + Ara-C
Number analyzed (Participants) | 1 | 3 | 5 | 4 | 18 | 3
h*ng/mL | 671 | 809 (439) | 1550 (484) | 3060 (1340) | 3840 (1520) | 8370 (2260)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were assessed at all study visits throughout the study from completion of Informed Consent Form (ICF) until End of Study for each patient, which is approximately 3 years
Groups:
- BL-8040 + Ara-C - All Patients: BL-8040 administration over two days followed by concurrent administration of BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days
- Open Label 2.0 mg/kg Period 6: BL-8040 2.0mg/kg + Ara-C: 2.0 mg/kg BL-8040 administration over two days followed by concurrent administration of 2.0 mg/kg BL-8040 with cytarabine (Ara-C) 1.5 or 3 g/m2/d per dose (based on age) over 5 days
Arm/Group | BL-8040 + Ara-C - All Patients | Period 1: BL-8040 0.5 mg/kg + Ara-C | Period 2: BL-8040 0.75 mg/kg + Ara-C | Period 3: BL-8040 1.0 mg/kg + Ara-C | Period 4: BL-8040 1.25 mg/kg + Ara-C | Period 5 & Expansion: BL-8040 1.5 mg/kg + Ara-C | Open Label 2.0 mg/kg Period 6: BL-8040 2.0mg/kg + Ara-C
All-Cause Mortality (participants affected / at risk) | 2/42 | 0/3 | 0/3 | 1/6 | 1/4 | 0/23 | 0/3
Serious Adverse Events (participants affected / at risk) | 21/42 | 1/3 | 3/3 | 3/6 | 1/4 | 10/23 | 3/3
Other Adverse Events (participants affected / at risk) | 41/42 | 3/3 | 3/3 | 6/6 | 4/4 | 22/23 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BL-8040 + Ara-C - All Patients (N=42) | Period 1: BL-8040 0.5 mg/kg + Ara-C (N=3) | Period 2: BL-8040 0.75 mg/kg + Ara-C (N=3) | Period 3: BL-8040 1.0 mg/kg + Ara-C (N=6) | Period 4: BL-8040 1.25 mg/kg + Ara-C (N=4) | Period 5 & Expansion: BL-8040 1.5 mg/kg + Ara-C (N=23) | Open Label 2.0 mg/kg Period 6: BL-8040 2.0mg/kg + Ara-C (N=3)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 11 (11) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 6 (6) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — HYPERSENSITIVITY
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE FEBRILE NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BL-8040 + Ara-C - All Patients (N=42) | Period 1: BL-8040 0.5 mg/kg + Ara-C (N=3) | Period 2: BL-8040 0.75 mg/kg + Ara-C (N=3) | Period 3: BL-8040 1.0 mg/kg + Ara-C (N=6) | Period 4: BL-8040 1.25 mg/kg + Ara-C (N=4) | Period 5 & Expansion: BL-8040 1.5 mg/kg + Ara-C (N=23) | Open Label 2.0 mg/kg Period 6: BL-8040 2.0mg/kg + Ara-C (N=3)
INJECTION SITE REACTION (General disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 9 (10) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (15) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 9 (10) | 0 (0)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 7 (7) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 17 (18) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 10 (10) | 1 (2)
Gingival bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 16 (20) | 2 (2) | 1 (2) | 3 (3) | 1 (1) | 7 (10) | 2 (2)
Vomiting (Gastrointestinal disorders) | 13 (15) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 9 (10) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukoplakia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 11 (11) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 9 (9) | 0 (0)
Pyrexia (General disorders) | 9 (11) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (9) | 0 (0)
Chills (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 11 (12) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site joint pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 25 (55) | 1 (1) | 3 (3) | 4 (9) | 2 (2) | 13 (36) | 2 (4)
Injection site pruritus (General disorders) | 10 (11) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 6 (7) | 0 (0)
Injection site rash (General disorders) | 11 (11) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
Injection site swelling (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Generalised oedema (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Chest pain (General disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Enterococcal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Enterobacter test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglicaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 10 (11) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 8 (9) | 0 (0)
Headache (Nervous system disorders) | 15 (17) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 7 (9) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (10) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 13 (13) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 7 (7) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 7 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Hypertension (Vascular disorders) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Flushing (Vascular disorders) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-03-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT01838395/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT01838395/SAP_001.pdf